CLINICAL TRIAL: NCT01787773
Title: VERITAS: An Evaluation of the Veniti Vidi Retrievable Inferior Vena Cava Filter System in Patients at Risk for Pulmonary Embolism
Acronym: VERITAS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IDE was withdrawn. Veniti no longer owns the rights to this device.
Sponsor: Veniti (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FIL-HUM-002P; ACTRN12612001255875 (Other: Australian New Zealand Clinical Trials Registry)
Record Dates: First submitted 2013-02-06; First posted 2013-02-11 (Estimated); Last update posted 2018-10-03 (Actual); Status verified 2018-10

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolus
Keywords: Inferior Vena Cava Filter; Vena Cava Filters
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Veniti Inferior Vena Cava Filter (Experimental)
  Interventions: Device: Veniti Inferior Vena Cava Filter

INTERVENTIONS:
Device: Veniti Inferior Vena Cava Filter

SUMMARY:
This is a prospective, multicenter single arm, nonrandomized study that will include 150 patients at a maximum of 20 investigational sites. It is estimated that it may take 13 months to complete enrollment. Follow-up will continue through 24 months post-implant or one month post-retrieval, whichever occurs first. It is required that filters be retrieved from at least 50 patients and the filter is permanent in at least 50 patients.

DETAILED DESCRIPTION:
Verify the effectiveness and safety of the Veniti IVC Filter in accordance with the clinical guidelines published by the Society for Interventional Radiology (SIR) .

The endpoint is clinical success (versus failure) at 6 months after implant or 1 month post retrieval, whichever occurs first, based on the definition provided by the SIR guidelines, as the absence of:

1. Procedure failure (assessed at the end of the implant procedure)
2. Subsequent pulmonary embolus
3. IVC occlusion
4. Filter embolization

Secondary assessments include:

Estimating the rate of:

1. Retrieval success
2. Device and procedure related adverse events
3. Assessing filter performance rate:

c1.Filter migration c2.Filter fracture c3.Filter Tilt

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Investigator judges caval filtration clinically indicated for prevention of pulmonary embolism in patient with venous thromboembolic disease or at high risk for venous thromboembolic disease. Patient must meet at least one of the following:
* Anticoagulant therapy is contraindicated, has failed, cannot be achieved or maintained, must be interrupted, resulted in complication, or places the patient at high risk of complication and the patient has:
* Pulmonary embolus
* Iliocaval deep vein thrombosis (DVT)
* Severe trauma with high risk of venous thromboembolism including closed head injury, spinal cord injury, or multiple long bone or pelvic fractures
* Surgery planned with high risk of venous thromboembolism including procedures such as bariatric, orthopedic, or pelvic surgery
* Past history of thromboembolic disease undergoing surgery

Therapeutic anticoagulation can be achieved, but the patient has:

* Venous thromboembolism such as pulmonary embolism or DVT with limited cardiopulmonary reserve
* Massive pulmonary embolism already treated with thrombectomy or any thrombolytic therapy
* Chronic pulmonary embolism already treated with thrombectomy
* Large, free floating proximal, e.g., iliofemoral or iliocaval, DVT
* Iliocaval DVT with planned catheter thrombectomy or thrombolysis treatment OR
* Medical condition with high risk of venous thromboembolism

Exclusion Criteria:

* Condition that inhibits radiographic visualization of the IVC
* Known inadequate venous anatomy to allow insertion or retrieval of the filter from the IVC including occlusion of the SVC or jugular veins
* Known IVC transverse diameter at target implant site > 28 mm
* Known obstructing abdominal mass or anatomy that is not suitable for infra-renal placement of IVC filter
* Known duplication of IVC or left-sided IVC
* Severe kyphosis or scoliosis
* Known IVC thrombosis extending to renal veins, or renal or gonadal vein thrombosis
* Risk for septic pulmonary embolism
* Confirmed bacteremia
* Estimated Glomerular Filtration Rate (eGFR) < 30 ml/min, or dialysis dependent.
* Contrast agent allergy that cannot be adequately pre-medicated
* Known hypersensitivity to Nitinol (nickel-titanium), platinum, Polyether ether ketone (PEEK), UV Cure Adhesive or Cyanoacrylate Adhesive
* Uncontrolled or active coagulopathy or known uncorrectable bleeding diathesis
* Life expectance < 6 months
* Female of childbearing potential who is pregnant or plans to become pregnant during the duration of the clinical study. (If a female of child bearing potential wishes to participate, she must have negative pregnancy test within 48 hours of the implantation and any retrieval procedures.)
* Has filter in place or underwent filter retrieval in previous 60 days
* Simultaneously participating in another therapeutic drug or device clinical trial or has participated in such trial in the 30 days prior to enrollment
* Investigator considers patient to be a poor candidate for the study or that including the patient may compromise the study, e.g., suspect patient may not comply with follow up procedures, concomitant conditions
* Patient does not wish to consent to study or comply with study procedures, including possible 2 year follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-03 (Estimated); Primary Completion 2015-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Success | 6 months
  The endpoint is clinical success (versus failure) at 6 months after implant or 1 month post retrieval, whichever occurs first, based on the definition provided by the SIR guidelines, as the absence of:
  * Procedure failure (assessed at the end of the implant procedure)
  * Subsequent pulmonary embolus
  * IVC occlusion
  * Filter embolization

SECONDARY OUTCOMES:
Secondary Endpoint | 24 months
  Estimating the rate of:
  * Retrieval success
  * Device and procedure related adverse events
filter performance rate | 24 months
  Assessing filter performance rate:
  * Filter migration
  * Filter fracture
  * Filter Tilt

CONTACTS AND LOCATIONS:
Locations (2):
- Alfred Hospital, Melbourne, Australia
- Auckland City Hospital, Grafton, New Zealand